CLINICAL TRIAL: NCT01567592
Title: Clinical Trial Evaluating the Treatment of Patients With Refractory Angina Pectoris With Low Intensity Extracorporeal Shockwave Therapy Device
Brief Title: Extracorporeal Shockwave Therapy for the Treatment of Chronic Angina Pectoris
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: Medispec (Industry)
Collaborators: KMH Cardiology and Diagnostic Centres (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESMR-KMH-Canada
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Refractory Angina Pectoris
Keywords: Extracorporeal Shockwave Therapy; Myocardial Ischemia; Refractory Angina
MeSH Terms: conditions — Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Shockwave Therapy (Experimental): Treatment group. Patients in this group receive actual shockwave therapy.
  Interventions: Device: Cardiac Extracorporeal Shockwave Therapy generator (Cardiospec)

INTERVENTIONS:
Device: Cardiac Extracorporeal Shockwave Therapy generator (Cardiospec) — Energy Density - 0.09 mJ/mm2
  Other Names: Cardiospec; ESMR therapy; Extracorporeal Shockwave Myocardial Revascularization

SUMMARY:
Low intensity shockwaves have been proven in animal studies to induce local growth of new blood vessels from existing ones.

The hypothesis of this study is that shockwave therapy could improve the symptoms of patients with refractory angina not amenable to revascularization with angioplasty or bypass surgery.

DETAILED DESCRIPTION:
Low intensity shockwaves (1/10 the ones used in Lithotripsy) are delivered to myocardial ischemic tissue. Shockwaves are created by a special generator and are focused using a shockwave applicator device. The treatment is guided by standard echocardiography equipment. The shockwaves are delivered in synchronization with Patient R-wave to avoid arrhythmias. The treatment is painless.

At first, the patient undergoes stress- SPECT testing to identify the ischemic areas. Following that, the same area is localized by the ultra-sound device and the shockwaves are focused to the ischemic area. Several treatments are required for optimal results.

ELIGIBILITY:
Inclusion Criteria

1. The patient will have an acoustic window to the myocardium by echocardiography. 4 chamber view (4CH), 2 chamber view (2CH), long axis (LAX) and short axis view (SAX) should be verified.
2. Patient is diagnosed with chronic angina pectoris. Diagnosis is based on medical history, complete physical evaluation, and Exercise SPECT.
3. Patient has documented myocardial reversible ischemia and or hibernation in at least one segment.
4. Patient is classified as AP CCS of III or IV.
5. Patient should be on a stable dosage of medication used to treat angina for at least 6 weeks prior to enrollment.
6. Patients demonstrates exercise tolerance time (ETT) duration < 10 minutes on a modified Bruce protocol on 2 consecutive tests (tests no less than 24 hours and no more than 2 weeks apart), with the second test within the difference of 25% of the first (Patients should not be informed of exercise restrictions required for entry into the study).
7. Patients where angioplasty and bypass are not indicated because of anatomical or procedural reasons or frequent reocclusion/restenosis following traditional revascularization.
8. Patient has refused to undergo another angioplasty or CABG.
9. Patient has signed an informed consent form.
10. Patient's condition should be stable and should have a life expectancy of > 12 months.
11. Patient's current and past medical condition and status will be assessed using previous medical history, physical evaluation, and the physicians (principle investigator's) medical opinion.

Exclusion Criteria

1. Patient has chronic lung disease based on the GOLD criteria the patient has stage IV: Very Severe COPD according to Spirometric Classification of COPD, Severity based on Post-Bronchodilator
2. Patient has emphysema and pulmonary fibrosis.
3. Patient has active endocarditis, myocarditis or pericarditis.
4. Patient is simultaneously participating in another device or drug study, or has participated in any clinical trial involving an experimental device or drug, including other drugs or devices enhancing cardiac neovascularization, or was treated with TMR (Transmyocardial revascularization) or PMR (Percutaneous revascularization) , or any ESWT machine for neovascularization of a competitor company within 3 months of entry into the study.
5. Patients who are unwilling or unable to cooperate with study procedure.
6. Patients who are unwilling to quit smoking during the study procedure (including screening phase)
7. Patients who had MI less than 3 months prior to treatment
8. Patients with moderately severe or severe valvular disease. Moderately-severe and severe disease will be echographically diagnosed as follows:

   * Aortic Stenosis: Patients with Moderately-severe [Peak Aortic valve gradient (AVG): 50-60 mmHg; Mean AVG: 30-40 mmHg; Effective orifice area (EOA): 0.75-1.0 cm2] and severe Aortic Stenosis [Peak AVG: above 60 mmHg; Mean AVG: above 40 mmHg; EOA: below 0.75 cm2]
   * Mitral Stenosis: Patients with severe Mitral Stenosis [EOA: below 1 cm2; Pressure half-time (ms): above 200 mmHg; Mean Mitral valve gradient: above 10 mmHg]
   * Aortic Regurgitation & Mitral Regurgitation: Patients with moderately- severe and severe aortic regurgitation and mitral regurgitation will be excluded.
   * Moderately-severe (grade 3, or 3/4) and severe (grade 4, or 4/4) are hemodynamically significant.
   * Tricuspid Regurgitation (TR): Its severity is graded from 1-4 as for aortic and mitral regurgitation. Grades 3 and 4 will be excluded from the study. The more severe levels of TR are common in severe biventricular failure, mitral stenosis, cor pulmunale and any other cause of pulmonary hypertension.
9. Patient with intraventricular thrombus
10. Patient is pregnant
11. Patient with a malignancy in the area of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Time to Angina | 6 months
  Change in time to angina using the modified Bruce exercise test from baseline to the 6 moths post baseline assessment

SECONDARY OUTCOMES:
Change in SPECT | 6 months
  The change in perfusion in pharmacological induced stress SPECT test (at rest and at stress) from baseline to 6 months post baseline (17 segments model).
Change in AP-CCS | 6 months
  The AP CCS Stage at the 6 months post baseline.
Total Exercise time | 6 months
  The change in Total Exercise Time (ETT) from baseline to 6 months post baseline.
Number of angina attacks (patient diary) | 6 months
  The change in the number of angina attacks from baseline to 6 months post baseline. The number of attacks per week will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Arvi Grover, MD, Principal Investigator — KMH Cardiology & Diagnostic Centers
Locations (1):
- KMH Cardiology & Diagnostic Centers, Ontario, Canada